CLINICAL TRIAL: NCT06543238
Title: The Effect of Breastfeeding Education Using the Card Game Method on Breastfeeding Success, Breastfeeding Self-efficacy and Satisfaction in Primiparous Mothers: A Randomized Controlled Trial
Brief Title: Breastfeeding Education Using the Card Game Method
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Sakine Yılmaz, Assistant Professor Doctor, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CakırıKU
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Primiparity
Keywords: Primiparity; Mothers; Breast Feeding; Self Efficacy; Education; Game
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The study consists of two groups: control and experimental group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Since the application will be performed by the researcher, patients will be blinded in this study. The statistician will be blinded in the evaluation of the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breastfeeding card game (Experimental): Breastfeeding card game group: Breastfeeding education will be given to 30 primiparous pregnant women in the intervention group using the card game method twice, two weeks apart.
  Interventions: Other: Breastfeeding card game group
- Control Group (No Intervention): No application will be made to this group by the researcher.

INTERVENTIONS:
Other: Breastfeeding card game group — Breastfeeding card game group: Breastfeeding education will be given to 30 primiparous pregnant women in the intervention group using the card game method twice, two weeks apart.
  Arms: Breastfeeding card game

SUMMARY:
This study aims to determine the effects of breastfeeding education using the card game method on breastfeeding success and breastfeeding self-efficacy in primiparous breastfeeding mothers.

DETAILED DESCRIPTION:
Breastfeeding is a safe feeding method that meets all nutritional and health needs of infants, strengthens immunity, protects against invisible microbes such as diarrhea and pneumonia, and improves growth, development, health and survival. Exclusive breastfeeding for 6 months and continuing breastfeeding for 2 years can improve the physical, mental and emotional health of mothers and their babies.

The World Health Organization recommends exclusive breastfeeding for up to 6 months and breastfeeding with complementary feeding until 2 years of age and beyond, as it is directly related to improving health and preventing infant morbidity and mortality. Problems that cause mothers not to breastfeed exclusively include lack of knowledge about the benefits of breastfeeding, proper breastfeeding, lack of breastfeeding consultancy services and support from health professionals, socio-cultural perceptions against breastfeeding, and lack of motivation to breastfeed.The development and implementation of effective training programs to improve breastfeeding self-efficacy is an important issue for health professionals.Therefore, the implementation of innovative strategies and methods in the field of health education can greatly contribute to women's learning in order to strengthen participation in preventive behaviors and promote breastfeeding.One of these educational methods is the card game method. Health messages are presented in various game formats such as four-card games. The educational and teaching method that uses a specific set of cards with various pictures, words and categories is a game. Card games are fun and educational games. This method has the advantages of being simple, being playable anywhere, being easy to store, being able to be played by children or adults in large or small groups and the participants being able to actively participate in the game.Nurses, who are the basic building blocks of health services, also need to provide effective care that is appropriate for the needs of the age. In this context, the educational approaches used by nurses are important. In nursing education, the use of game-based learning and teaching methods has attracted attention, especially in recent years. Game-based learning, one of the educational methods, has an important effect in increasing individuals' interest in educational subjects, ensuring the permanence of knowledge and creating motivation.It is important for health professionals to provide training and consultancy to women on this issue in order to manage the breastfeeding process correctly, which is important for the health of both the mother and the baby. In this direction, as a result of this study, it is thought that by creating special breastfeeding cards and using a gamification-based education model, correct breastfeeding behavior and self-sufficiency will be developed in mothers. No study has been found in our country where this method has been used. In this respect, the study is original. As a result of the study, it is thought that the use of this game education model by health professionals while providing breastfeeding education and consultancy will facilitate the breastfeeding process.

ELIGIBILITY:
Inclusion Criteria:

* The conditions for volunteering to participate in the study are being over the age of 18, being able to read and write, being able to read and understand Turkish, not having hearing, speaking or visual impairments, having received breastfeeding training at a pregnancy school, being healthy in the 34th to 38th week of primiparous pregnancy, having a planned cesarean section, having a live birth and having a healthy baby.

Exclusion Criteria:

* Obstacles to communication include having a visual, hearing or perception disorder, not being able to read or write, having a psychiatric illness, being multiparous and having a vaginal birth, having a risky pregnancy, not having a live birth and not having a live baby after birth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since it is a study conducted on pregnant women, it concerns the female gender.
Enrollment: 60 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale | 36th week of pregnancy and postpartum
  The scale consists of a total of 14 items that evaluate breastfeeding self-efficacy. The scale is a 5-point Likert-type scale, and the items are evaluated by rating from 1 = "not sure at all" to 5 = "always sure". The lowest score that can be obtained from the scale is 14, the highest score is 70; higher scores indicate higher breastfeeding self-efficacy.

SECONDARY OUTCOMES:
LATCH Breastfeeding Diagnostic and Assessment Scale | It will be applied to women in the control and experimental groups after birth.
  LATCH focuses on 5 features to be able to take appropriate action in cases where intervention is necessary for the mother. L (Latch): Baby's latching on to the breast, A (Audible Swallowing): Baby's swallowing sound is heard, T (Type of Nipple): Type of nipple, C (Comfort of Breast/Nipple): Mother's comfort with the breast/nipple H (Hold/Position): Defined as the assistance the mother needs to place her baby in the breastfeeding position. Each of the criteria is evaluated as "0, 1, 2" points. The maximum score that can be obtained is 10, and a high score from the evaluation and diagnosis scale means that breastfeeding success is high.
Visual analog satisfaction scale | It will be applied to women in experimental groups after birth.
  It is a scale used to evaluate satisfaction with the training provided. The individual indicates his/her satisfaction by marking a score between 0 (not satisfied at all) and 10 (very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Sakine Yılmaz, Principal Investigator — Çankırı Karatekin University
Locations (1):
- Sakine Yılmaz, Çankırı, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No